CLINICAL TRIAL: NCT07236671
Title: International Multi-centre, Prospective, Longitudinal Cohort to Evaluate the Progression Pattern of Choroidal Venous Alterations
Brief Title: Progression Patterns of Choroidal Venous Alterations
Acronym: CVA
Status: Recruiting | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National University Hospital, Singapore (Other); University of Malaya (Other); Hong Kong University (Other)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore National Eye Centre
Other Study IDs: 2024-4359
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pachychoroid Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is about understanding how a condition called pachychoroid changes over time. Pachychoroid refers to an anatomic choroidal characteristic with abnormally thick choroid or abnormally dilated Haller's vessels. Pachychoroid can range from mild forms which does not cause any problems to more serious ones that might cause vision loss.This study will recruit participants with pachychoroid, to learn more about how this condition develops, how it affects people in the long run, and what factors might make it worse.

DETAILED DESCRIPTION:
This study aims to document the longitudinal progression pattern and the incidence rate of progression of choroidal venous alteration (defined as either an increase in number of quadrants with pachyvessels or formation of new anastomoses which violates the physiological watershed It will provide valuable natural history data to study the pattern of evolution of choroidal vessels over time and validate the proposed multi-hit theory over a period of three years.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 45 years or older.
2. Presence of pachyvessels on ultra-widefield (UWF) imaging in at least one quadrant.
3. Willing to undergo pupil dilation, and protocol-required procedures for both eyes
4. Willing to provide written informed consent

Exclusion Criteria:

1. Presence of disorders of the ocular media which interfere with visual acuity and other ocular assessments during the study period
2. Eyes with other ocular pathology such as trauma, inflammation, previous intraocular surgery (except for cataract surgery)
3. Systemic diseases that might affect ocular blood flow such as uncontrolled hypertension, autoimmune disease, and haematological disorders
4. Pregnant or nursing women
5. Persons who are unable to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will aim to recruit 170 participants in Singapore National Eye Centre (SNEC) and 50 participants in National University Hospital, 30 participants from the University of Malaya
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Progression of choroidal venous alterations | 3 years
  Proportion of eyes demonstrating progression of choroidal venous alterations, defined as either an increase in number of quadrants with pachyvessels or formation of new choroidal anastomoses.

SECONDARY OUTCOMES:
Incidence of progression of pachychoroid disease manifestation | 3 years
  New onset of Central Serous Chorioretinopathy (CSCR), focal Retinal Pigment Epithelium (RPE) changes, or other pachychorois related findings.
Risk factors associated with progression of choroidal venous alteration | 3 years
  Assessment of demographic, cilinical, and imaging parameters associated with progression.

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong University, Hong Kong, Hong Kong
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Singapore National Eye Centre/ Singapore Eye Research Institute, Singapore

IPD SHARING:
Plan to Share IPD: No